CLINICAL TRIAL: NCT02211378
Title: Effects of Stress on Observers and Their Subsequent Performance During High Fidelity Simulation-based Training: A Randomized Controlled Trial.
Brief Title: Effects of Stress on Observers and Their Subsequent Performance During High Fidelity Simulation-based Training.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: KK Women's and Children's Hospital (Other Government)
Collaborators: Singhealth Foundation (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: None
Other Study IDs: CIRB2012/402/D
Record Dates: First submitted 2014-08-05; First posted 2014-08-07 (Estimated); Last update posted 2014-08-07 (Estimated); Status verified 2014-08

CONDITIONS: Stress
Keywords: stress; performance; cortisol
MeSH Terms: interventions — Observer Variation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Observer (Experimental): Trainees are in the role of observers (not actively participating in simulation scenario) during first 2 simulation sessions, then placed in the role in the 'hotseat' actively participating during the third simulation session.
  Interventions: Other: Observer
- Hotseat (Active Comparator): Trainees are in the 'hotseat' actively participating during all 3 simulation sessions
  Interventions: Other: Hotseat

INTERVENTIONS:
Other: Observer — Trainees are in the role of observers (not actively participating in simulation scenario) during first 2 simulation sessions, then placed in the role in the 'hotseat' actively participating during the third simulation session.
  Arms: Observer
Other: Hotseat — Trainees in the hotseat group are placed in the 'hotseat' to actively participate and manage the simulated medical crises in the simulation scenarios.
  Arms: Hotseat

SUMMARY:
This randomized controlled trial aims to determine if the stress response and performance of trainees who are observers in simulation training is similar to trainees who are actively participating in simulation training in the 'hotseat' during 3 consecutive simulation sessions.

We hypothesize that trainees experience less stress when they are observers in the first 2 simulation sessions. However, when they are placed in the 'hotseat' during the third session, their stress response, as well as their performance, will be similar to trainees who spend all 3 simulation sessions in the 'hotseat'.

DETAILED DESCRIPTION:
Background: High fidelity simulation-based training (SBT) using sophisticated manikins instead of real patients for medical teaching is now commonly practiced worldwide. We previously showed that SBT causes significant stress in the trainees, as evidenced by a rise in their heart rate and salivary cortisol(; and that repeated exposure to SBT was associated with the same level of stress, despite performance improving. From our studies, participants in the 'hot-seat' actively managing the clinical crisis experience the highest levels of stress but benefit the most from the learning experience. However, the stress experienced by observers (who are in the same room but not actively managing the crisis) and their learning outcomes have not been studied.

Objectives: We aim to determine: 1) If observers of SBT experience less stress when compared to the trainees in the 'hot-seat' and; 2) if trainees who were observers in prior SBT sessions perform as well as trainees who were in the 'hot-seat' during subsequent SBT sessions.

Methodology: Thirty-six trainee anaesthetists are randomized into 2 groups to undergo three SBT scenarios. 18 Trainees randomized to the Observer group will first undergo two SBT scenarios as observers followed by a third session in the 'hot-seat'. 18 Trainees in the Control group will undergo all 3 sessions in the 'hot seat'. For each session, stress response is measured by salivary cortisol and amylase while performance is measured using the Anaesthetists Non Technical Skills (ANTS) score.

Clinical Significance: If we find that trainees who are observers of the first 2 SBT scenarios experience less stress than the 'hot-seat' trainees but yet achieve similar level of performance during the third SBT session, we can potentially make SBT less stressful and reduce the total number of simulation required, thus improving the efficiency of simulation training.

ELIGIBILITY:
Inclusion Criteria:

* Anaesthesia residents in their 2nd or 3rd year of training

Exclusion Criteria:

* Hypertension
* Cardiac disease
* Endocrine disorder
* Use of beta-blockers
* Recent stressful or traumatic life events
* Pregnancy

Ages: 24 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 33 (Actual)
Dates: Start 2012-09; Primary Completion 2014-02 (Actual); Study Completion 2014-02 (Actual)

PRIMARY OUTCOMES:
Change in Salivary Cortisol from baseline | From baseline to end of the simulation session, typically after 15 minutes.
  Salivary cortisol measurement. Saliva collected using Salimetric oral swabs and salivary cortisol measured using ELISA technique.

SECONDARY OUTCOMES:
Salivary amylase | From baseline to end of the simulation session, typically after 15 minutes.
  Saliva collected using Salimetric oral swabs and analyzed using ELISA technique
Anaesthetist's non-technical skills score | During simulation, typically lasting 15 minutes.
  Anaesthetist's non-technical skills score: a validated and reliable marking system measuring non-technical skills comprising 4 elements including task management, teamwork, situation awareness and decision making.
DASS questionnaire | At the end of simulation session
  Subject's self assessment of stress using the Depression, Anxiety and Stress questionnaire

CONTACTS AND LOCATIONS:
Overall Officials: Choon L Bong, MBChB FRCA, Principal Investigator — KK Women's and Children's Hospital, Singapore
Locations (1):
- KK Women's and Children's Hospital, Singapore, Singapore, Singapore

REFERENCES:
- [Background] Bong CL, Lightdale JR, Fredette ME, Weinstock P. Effects of simulation versus traditional tutorial-based training on physiologic stress levels among clinicians: a pilot study. Simul Healthc. 2010 Oct;5(5):272-8. doi: 10.1097/SIH.0b013e3181e98b29. PMID 21330809
- [Derived] Bong CL, Lee S, Ng ASB, Allen JC, Lim EHL, Vidyarthi A. The effects of active (hot-seat) versus observer roles during simulation-based training on stress levels and non-technical performance: a randomized trial. Adv Simul (Lond). 2017 Mar 20;2:7. doi: 10.1186/s41077-017-0040-7. eCollection 2017. PMID 29450008